CLINICAL TRIAL: NCT05487534
Title: Impact of Glycemic Variability on Cognitive Impairment, Disordered Eating Behavior, and Self-management Skills in Patients Living with Type 1 Diabetes
Brief Title: Do "sugar Swings" Impact the Brain Function and the Eating Behaviors of People with Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Collaborators: CHU de Quebec-Universite Laval (Other); Institut de Recherches Cliniques de Montreal (Other); Centre d'expertise Poids, Image et Alimentation (CEPIA) (Unknown); Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Sylvain Iceta, Principal Investigator, Laval University
Other Study IDs: MP-20-2023-6466
Record Dates: First submitted 2022-07-08; First posted 2022-08-04 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes; Cognition; Eating behaviors; Glycemic variation; Blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Feeding Behavior | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sugar Swing +: Patients with type 1 diabetes with a high glucose variability (i.e., a coefficient of variation > 36% over a 10-day continuous glucose monitoring)
  Interventions: Other: Observational
- Sugar Swing -: Patients with type 1 diabetes with low glucose variability (i.e., a coefficient of variation < 36% over a 10-day continuous glucose monitoring)
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — The same self-reported questionnaires and cognitive tests will be completed by both groups. There is no intervention.

SUMMARY:
In type 1 diabetes, it is common to choose the food we eat according to the blood sugar level and the insulin dose and vice versa. Beyond the nutritional aspects, the relationship to food and the resulting eating behaviors can be a source of suffering. Also, it has been reported that one out of two people over 60 years of age living with type 1 diabetes has cognitive impairment. Changes in cognitive functions can have important implications for daily well-being, diet (e.g., the ability to modulate cravings), and treatment decisions to manage diabetes.

One factor that can affect both eating behaviors and cognitive function is variation in blood glucose levels.

This research aims to better understand the impact of glycemic variability in disordered eating behaviors and cognitive impairment, and its consequences on self-management skills in people with type 1 diabetes.

The hypotheses are that i) higher glycemic variability is associated with higher disordered eating behaviors and poorer cognitive function in people with type 1 diabetes, and that differences exist between sexes, ii) higher disordered eating behaviors and poorer cognitive function are associated with lower self-management skills; and iii) cognitive impairment, interoception awareness and insulin resistance may mediate the relationship between glycemic variability and disordered eating behaviors.

This research study will contribute to highlighting the consequences of blood sugar fluctuations, "sugar swings", in daily life, in particular the way they disrupt eating behaviors and brain function. A better understanding of the mechanisms involved could eventually allow for early detection and management of these problems. Our study will also seek to understand the patients' point of view, which will allow the design of appropriate and meaningful recommendations.

DETAILED DESCRIPTION:
All assessments will be done in virtual mode through secure platforms (but also offered in person in Quebec City if needed to limit discrimination).

The study will start with an inclusion visit during which self-reported and medical data will be collected as well as some anthropometric parameters measured. Following the visit, the participant will be asked to wear a continuous glucose sensor provided by the investigator (Dexcom®) to perform a continuous glucose recording for 10 days. During this 10-day period, the participant will be required to complete:

* A food diary during 3 weekdays and 1 weekend day using the Keenoa® app.
* 3 online sessions combining questionnaires (using the Redcap platform) and computerized tests (Inquisit® platform). Each session will last approximately 45 minutes (can vary between 30 and 60 minutes).

Participants who wish to participate in the qualitative phase of this study will also be offered the opportunity to do so. Participants will be recruited consecutively until a total of 50 are reached. For this part of the study, an individual interview will be conducted by a professional specifically trained in this method of analysis. This meeting will last on average 1.5 hours, but may last up to 2.5 hours depending on the length of the discussion. There will be an audio and video recording of this meeting. The discussions will then be transcribed into text and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes (> 12 months)
* Age between 18 and 65 years old
* 6.5 % < A1C < 9% (to avoid potential severe eating disorder)

Exclusion Criteria:

* Type 2 diabetes or other form of diabetes; gastroparesis (clinical diagnosis);
* Recent (< 6 months) major cardiovascular event (e.g. myocardial infarction, cerebrovascular accident, major revascularization)
* Recent (< 12 weeks) severe hypoglycemia episodes (<2.8 mmol/L or assistance from a third party)
* Recent (< 12 weeks) changes in insulin type or delivery method
* Automated Insulin Delivery
* History of severe brain trauma, epilepsy, schizophrenia or bipolar disorders
* Inability to use a computer
* Incorrect vision or auditory problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited through the endocrinology clinics of the CHU de Québec (approximately 1000 patients living with type 1 diabetes) and the Institut de recherches cliniques de Montréal (IRCM) (>800 patients living with type 1 diabetes). We will also recruit through the BETTER registry, overseen by Dr. Rabasa-Lhoret and Dr. Brazeau (collaborators on the project) and co-funded by IRSC and JDRF: over 2000 people with type 1 diabetes are currently enrolled in the registry and 98% of participants have agreed to be contacted for future research studies. In case of recruitment difficulties, an announcement will also be made on social networks (such as Facebook).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder examination (EDE-Q) | Day 1 (+/- 2 days)
  To assess eating behaviors according to their glycemic variability.
Glucose variability and insulin resistance (CGMS - 10 days) | Start at inclusion (Day 1 to Day 10)
  CGMS will be performed over a 10-day period using a DEXCOM G6 to separate participants into groups based on glycemic variation (i.e., a coefficient of variation [CV] >36% over a 10-day CGMS) versus those with a low glucose variability (i.e., CV <36%).

SECONDARY OUTCOMES:
Distress Diabetes Scale (T1-DDS) | Inclusion
  To assess self-management's skills.
Diabetes Behavior Ratting Scale (DBRS) | Inclusion
  To assess self-management's skills.
Generalized Anxiety Disorder (GAD-7) | Inclusion
  To assess anxiety disorders.
Patient Health Questionnaire (PHQ-9) | Inclusion
  To assess depression disorder.
Diabetes Numeracy Test (DNT-15) | Inclusion
  To assess diabetes literacy and numeracy skills.
Physical and psychological comorbidities | Inclusion (medical data)
  Including eating disorders.
Diabetes Information : Duration | Inclusion (medical data)
  Number of years since the diagnosis of diabetes.
Diabetes Information : Modality of insulin delivery | Inclusion (medical data)
  Pumps or injections of insulin.
Diabetes Information : Total daily insulin dose | Inclusion (medical data)
  The dose of insulin taken per day.
Diabetes Information : Duration of diabetes self-monitoring | Inclusion (medical data)
  Number of years or months of its use, either self-monitoring with capillary glucose tests or CGMS.
Diabetes Information : Severe hypoglycemic episodes | Inclusion (medical data)
  Number of severe hypoglycemic episodes over the last year.
Diabetes Information : Medication | Inclusion (medical data)
  Past year and current medications (included use of psychotropic drugs to be considered as a potential confounding factor).
Diabetes Information : Diabetes complications | Inclusion (medical data)
  Number and type of diabetes complications.
Diabetes Information : Coefficient of variation | Inclusion (medical data)
  Measured coefficient of variation based on previous CGMS and last available HbA1c (max 6 months).
Anthropometric markers : BMI | Inclusion (medical data)
  Weight and height will be combined to report BMI in kg/m^2.
Anthropometric markers : Waist, hips and neck circumferences | Inclusion (medical data)
  Waist, hips and neck circumferences will be self measured in cm with a measuring tape.
Biological information : Cholesterol and triglycerides | Inclusion (biological data)
  Measurement of cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides in mg/dL.
Biological information : Fasting blood glucose | Inclusion (biological data)
  Measurement of fasting blood glucose in mg/dL.
Biological information : C-peptide | Inclusion (biological data)
  Measurement of c-peptide in nmol/L.
Biological information : Triglycerides | Inclusion (biological data)
  otal cholesterol, triglycerides, HDL-cholesterol, LDL-cholesterol, fasting blood glucose, c-peptide, ghrelin fasting and CRP
Biological information : Ghrelin fasting and C-Reactive protein (CRP) | Inclusion (biological data)
  Measurement of ghrelin fasting and CRP in mg/L.
Detail and Flexibility Questionnaire (DFQ) | Day 1 (+/- 2 days)
  To assess cognitive flexibility.
Adult ADHD Self-Report Scale (ASRS) | Day 1 (+/- 2 days)
  To screen for Attention Deficit Hyperactive Disorder (ADHD).
Category Switch Task | Day 1 (+/- 2 days)
  To assess attention.
Multidimensional Assessment of Interoceptive Awareness Version 2 (MAIA) | Day 4 (+/- 2 days)
  To assess the level of interoception.
Binge Eating Scale (BES) | Day 4 (+/- 2 days)
  To assess eating behaviors.
Tower of London Task | Day 4 (+/- 2 days)
  To assess executive functioning.
Stop Signal Task | Day 4 (+/- 2 days)
  To assess impulsivity and inhibition.
5-Trial Adjusting Delay Discounting | Day 4 (+/- 2 days)
  To assess temporal discounting.
Short UPPS-P Impulsive Behavior Scale | Day 8 (+/- 2 days)
  To assess behavior impulsivity.
Modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) | Day 8 (+/- 2 days)
  To estimate susceptibility to food reward.
Emotional Go/No-Go Task | Day 8 (+/- 2 days)
  To assess inhibition leverages by emotion recognition and regulation.
Attentional Cueing Procedure | Day 8 (+/- 2 days)
  To assess the effects of threat stimuli on capturing and holding attention.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Iceta, MD, PhD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (2):
- Canada (2):
  - IRCM, Montreal
  - CHU de Québec, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Iceta S, Sohier L, Begin C, Brazeau AS, Rabasa-Lhoret R, Gagnon C. Impact of glycemic variability on cognitive impairment, disordered eating behaviors and self-management skills in patients with type 1 diabetes: study protocol for a cross-sectional online study, the Sugar Swing study. BMC Endocr Disord. 2022 Nov 18;22(1):283. doi: 10.1186/s12902-022-01191-4. PMID 36401237